CLINICAL TRIAL: NCT05040997
Title: Small Airways Disease (SAD) in Severe Asthma as a Novel Endpoint and Distinct
Brief Title: Small Airways Disease (SAD) in Severe Asthma as a Novel Endpoint and Distinct Target for Mepolizumab (SASAM Study)
Acronym: SASAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3999
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Small Airway Disease; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Small airways assessment — Small airways assessment

SUMMARY:
Rationale Although the majority of asthma patients can be effectively treated with currently available medications, a substantial subset remains severe, causing a considerable proportion of resource expenditure. Severe asthma is now widely accepted to be a heterogeneous syndrome consisting of multiple phenotypes identified by specific biomarkers and targeted by tailored biological therapies. However, much remains unclear regarding the best approaches to manage these patients, or concerning the pathophysiological mechanisms underlying the disease.

Small airways (SA) are defined as those airways with an internal diameter <2 mm. In patients affected by asthma, it has been reported that SA are the predominant site of airflow resistance. Peripheral airways are thickened in asthma due to chronic inflammation in the epithelium, submucosa and muscle area. It has been suggested that the outer wall is more inflamed than the inner wall, with a higher number of lymphocytes, eosinophils, and neutrophils associated to an increased mRNA expression of interleukin-4 (IL-4), IL-5 and eotaxin. Moreover, it is well documented that SA inflammation and dysfunction contributes significantly to the clinical impact of asthma and that 50-60% of asthmatics have a SA involvement across all disease severities. An important question is whether SA disease in asthma is variable among distinct asthma phenotypes and whether it occurs in all patients. Cluster analyses have been recently used to identify specific asthma phenotypes, but markers of SA function have not been investigated. However, evidence is accumulating to support the concept that SA dysfunction and inflammation may contribute to distinct asthma phenotypes. Recent findings indicate that SA are significantly affected in severe asthma and that their involvement is associated with worse disease outcomes. It has been reported that patients with asthma and a history of frequent exacerbations per year had a significant SA involvement Furthermore, peripheral airways significantly contribute not only to the level of asthma control, but also to patients' quality of life and perception of symptoms. At last more thickened SA and higher numbers of eosinophils are detectable in subjects with fatal asthma.

The assessment of SA represents a big challenge and requires qualified expertise and sophisticated techniques including body plethysmography, single and multiple breath nitrogen washout, impulse oscillometry (IOS), fraction exhaled NO at multiflow, sputum induction and high-resolution chest CT (HRCT). Such procedures can either provide functional information on the degree/extent of ventilation heterogeneity and air trapping or facilitate the understanding of the inflammatory and remodeling processes. These measures are not usually part of the evaluation of asthmatic patients and in the monitoring of the effects of drugs recommended for severe asthma.

Mepolizumab represents an innovative weapon for the treatment of severe eosinophilic asthma. In most of these patients the drug controls inflammation, improves lung function, ameliorates clinical symptoms, reduces exacerbations and has a marked steroid-sparing effect. However, there is still a significant proportion of non-responders and a lack of validated predictive biomarkers in such subpopulation. In regard to this, very limited findings are available about the effect of mepolizumab on SA. At the best of our knowledge, the only paper available in literature, addressing the topic, is the study of Farah and co-workers. The authors found that an early improvement in SA function was associated with better asthma control and represented a significant contributor to the therapeutic response. However, the study was conducted in a limited cohort of patients, assessing SA only through multi breath nitrogen washout, and not considering the relationship between SA disease and levels of peripheral/sputum eosinophils. Also, a study was recently initiated at the Hopitaux de Paris to evaluate airway remodelling during mepolizumab treatment (REMOMEPO, NCT03797404).

A better definition of severe asthma phenotypes and endotypes, as well as the identification of novel disease targets and biomarkers to predict treatment response and monitor efficacy and safety of biological drugs over time, would favor a Precision Medicine approach translating in both improved disease management and reduced healthcare costs and social burdens. This is considered a crucial unmet need and further research in the field is strongly recommended by international guidelines, respiratory scientific societies, healthcare systems and regulatory boards.

DETAILED DESCRIPTION:
Study hypothesis We hypothesize that mepolizumab has a significant beneficial effect on small airways disease in severe asthmatics and that the evaluation of small airways before and during treatment may represent a distinctive marker of response and a novel target for a preferential use of this drug vs other biologics available for severe eosinophilic asthmatic patients.

Study objectives

* To evaluate a wide panel of validated small airways endpoints in eosinophilic severe asthmatics before mepolizumab treatment
* To evaluate longitudinal changes of these endpoints at different time points during mepolizumab treatment
* To relate small airways endpoints recorded at baseline and their changes over time to other functional, laboratory, clinical and patient reported outcomes

Study center The study will be conducted at the Asthma Center of the Fondazione Policlinico Universitario A. Gemelli, IRCCS, Respiratory, Allergy and ENT Physicians closely and sinergically collaborate in the framework of the Asthma Center with shared clinical and research activities aimed to an optimal management of asthma and its comorbidities, as well as with regular meetings for multidisciplinary clinical case discussion and collective decisions on treatment strategies. The Asthma Center is part of the Italian Severe Asthma Network (SANI) and will be soon one of the coordinating centers for the newborn Italian Mild-Moderate Asthma Network (MANI), therefore representing a center of excellence and reference at a national level, with easy and wide access to the study population.

Study design Asthmatic patients referred to the Asthma Center and eligible for starting Mepolizumab, after having optimized adherence, inhalation technique and comorbidity management following multidisciplinary assessment, will enter a single-site oservational prospective longitudinal cohort study. Subjects will be monitored for 12 months and SA endpoints will be recorded at the beginning of the biological therapy (T0) and after 3,6,12 months (T3, T6, T12). SA endpoints will be also related to other functional, clinical and patient reported outcomes.

Study population Male and female subjects addressed to the Asthma Center, aged ≥12 yrs with severe asthma as defined by ATS/ERS guidelines (≥12months high-dose ICS + additional controller treatments), ≥2 exacerbations (corticosteroid and/or ED visit and/or hospitalization in the previous 12 months), blood eosinophil ≥150 cells/µl at study entrance or ≥300cells/µl historically and a smoking history <2 pack/year.

Study drug Mepolizumab 100mg via subcoutaneous administration

Study procedures

The following methodologies will be included in the study:

Clinical history, Demographics and questionnaires (i.e. ACT, ACQ, ACQLQ) Pulmonary function tests (i.e. spirometry, body plethysmography, single- and multi-breath nitrogen washout, impulse oscillometry) Airway inflammatory markers (i.e. fraction exhaled nitric oxide - FeNO) Allergy tests (i.e. skin-prick tests and immunoassays for total and specific serum IgE) Biological sampling (i.e. blood and sputum eosinophils)

Study endpoints The following endpoints relating to small airways involvement will be considered: R5, R20, X5, AX, RF, FEF25-75, TLC, RV, Raw, Gaw, DLCO, KCO, LCI

ELIGIBILITY:
Male and female subjects addressed to the Asthma Center, aged ≥12 yrs with severe asthma as defined by ATS/ERS guidelines (≥12months high-dose ICS + additional controller treatments), ≥2 exacerbations (corticosteroid and/or ED visit and/or hospitalization in the previous 12 months), blood eosinophil ≥150 cells/µl at study entrance or ≥300cells/µl historically and a smoking history <2 pack/year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects addressed to the Asthma Center, aged ≥12 yrs with severe asthma as defined by ATS/ERS guidelines (≥12months high-dose ICS + additional controller treatments), ≥2 exacerbations (corticosteroid and/or ED visit and/or hospitalization in the previous 12 months), blood eosinophil ≥150 cells/µl at study entrance or ≥300cells/µl historically and a smoking history <2 pack/year.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-09 (Estimated); Study Completion 2023-05-09 (Estimated)

PRIMARY OUTCOMES:
- To evaluate a wide panel of validated small airways endpoints in eosinophilic severe asthmatics before mepolizumab treatment | May 2023
- To evaluate longitudinal changes of these endpoints at different time points during mepolizumab treatment | May 2023
- To relate small airways endpoints recorded at baseline and their changes over time to other functional, laboratory, clinical and patient reported outcomes | May 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico universitario A. Gemelli - IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No